CLINICAL TRIAL: NCT05329636
Title: Fecal Auto-transplantation for Enteric Microbial Rehabilitation Post 14 Day Antibiotics Therapy Against Helicobacter Pylori Infection
Brief Title: Auto Fecal Microbial Transplant Post Helicobacter Pylori Antibiotic Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Shmuel Kivity, MD, director, R&D department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0278-18TLV
Record Dates: First submitted 2020-06-04; First posted 2022-04-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: FMT through capsules FMT through enema- open label in 3-4 patients to examine feasibility Control group without FMT
Who Masked: Participant, Investigator
Masking Description: Capsules will be either with FMT or placebo. Same appearance. Patients will be randomized to either arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo FMT capsules (Placebo Comparator): Glycerol and saline solution will be pipetted into commercially available acid-resistant hypromellose capsules (DRCaps, Capsugel) (650 μL), which will be closed and then secondarily sealed. Capsules will be stored frozen at -80°C (-112°F). Patients will swallow 30 frozen capsules on two consecutive days. Capsules look exactly the same as FMT capsules
  Interventions: Other: Placebo capsules
- FMT capsules (Experimental): Fecal matter solution (feces, glycerol and saline solution) will be pipetted into commercially available acid-resistant hypromellose capsules (DRCaps, Capsugel) (650 μL), which will be closed and then secondarily sealed. Capsules will be stored frozen at -80°C (-112°F). Patients will swallow 30 frozen capsules on two consecutive days.
  Interventions: Biological: Fecal Microbial Transplant (FMT)
- FMT enemas (Active Comparator): patients will evacuate the bowel prior to the procedure and will fast for 3 hours prior to the procedure . Patients will receive 80 ml of enema/ Fecal matter solution (feces(25 gr of stool , glycerol and saline solution) will be stored at 50 ml tubes frozen at -80°C (-112°F).
  Interventions: Biological: Auto Fecal Microbial Transplant (FMT) via enema

INTERVENTIONS:
Biological: Fecal Microbial Transplant (FMT) — FMT through capsules- patients will evacuate the bowel with 1 liter of Meroken solution 12 hours prior to the procedure and will fast from food for 12 hours prior to the procedure. Patients will swallow 30 frozen capsules on two consecutive days.
  Arms: FMT capsules
Other: Placebo capsules — Patients will evacuate the bowel with 1 liter of Meroken solution 12 hours prior to the procedure and will fast from food for 12 hours prior to the procedure. Patients will swallow 30 frozen placebo-capsules on two consecutive days.
  Arms: Placebo FMT capsules
Biological: Auto Fecal Microbial Transplant (FMT) via enema — 3.FMT through enema- patients will evacuate the bowel prior to the procedure and will fast for 3 hours prior to the procedure . Patients will receive 80 ml of enema. Enemas will be administered with the assistance of the study nurse. Patients will be asked to hold the enema content for at least 15 minutes.
  Arms: FMT enemas

SUMMARY:
Current guidelines mandate Helicobacter pylori (H. Pylori) eradication with 2-3 antibiotics for 14 days ,This may result in multiple side effects and in eradication of important bacterial species to human health, exposing humans to multiple disease conditions.

Preservation of fecal microbiome prior to antibiotic therapy and auto-transplantation of the microbes post H. pylori eradication, will enable avoiding eradication of beneficial microbial populations and perhaps protect from consequent disease conditions.

DETAILED DESCRIPTION:
This is a pilot study. Prior to antibiotics therapy for their baseline H.Pylori infection, patients will be asked to deliver at least 50 grams of fresh stool to the Tel Aviv Medical Center (TLVMC) Bacteriotherapy Clinic. All patients will receive therapy to eradicate H. Pylori according to current guidelines (14 days) and physician's discretion, and will be tested to validate H. pylori eradication, at least 21 days post therapy (according to guidelines: Kyoto/ ACG/ Maastricht). For patients that H. pylori was not eradicated- a second line therapy will be administered according to guidelines, and stool will be retrieved at an additional time point, before FMT and after successful H. pylori eradication.

Patients will be allocated into one of three groups:

1. Intervention group- patients will undergo Auto-FMT through capsules.
2. Intervention group-patients will undergo Auto-FMT through enema.
3. Control Group-patients will receive FMT through placebo capsules.

Patients in Intervention group will undergo an additional breath test for H. Pylori, 14-28 days post FMT, to exclude H. pylori-self infection, by the FMT. This concern is related to the capsules therapy, although the fecal filtrate is double packaged in two capsules (one inside another) which are designed to dissolve only in the duodenum at a basic pH.

If patients are found to be re-infected, they will undergo an additional antibiotics course and post eradication will receive FMT through an enema according to the above specified protocol.

FMT capsules will be generated at the laboratory of the Gastrointestinal department at the Tel Aviv Medical Center. The same procedure for FMT generation will be used in this study as in other studies of the IBD unit and in the clinical Bacteriotherapy setting.

FMT administration:

1. FMT through capsules (FMT/placebo)- patients will evacuate the bowel with 1 liter of Meroken solution 12 hours prior to the procedure and will fast from food for 12 hours prior to the procedure. Patients will swallow 30 frozen capsules on two consecutive days.
2. FMT through enema- patients will evacuate the bowel prior to the procedure and will fast for 3 hours prior to the procedure . Patients will receive 80 ml of enema. Enemas will be administered with the assistance of the study nurse. Patients will be asked to hold the enema content for at least 15 minutes.

At the post-FMT visit and follow -up visits, patients will be examined by a physician who will record clinical symptoms (abdominal pain, nausea, vomiting, weight change), adverse events (fever, abdominal pain, bloating, changes in bowel habits) and general well-being (quality of life and patient reported outcomes questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Positive H. pylori on either breath test or gastric biopsy
* Patient is intended to receive antibiotics therapy for H. pylori eradication

Exclusion Criteria:

* Severe systemic disease that may impact the microbiome. For example: heart disease, type two diabetes, chronic liver or kidney failure
* Antibiotics therapy during the prior 2 months to enrollment
* Planned to receive antibiotics within the upcoming 2 months (surgery etc) for reasons other than H. Pylori
* Inability to complete the study protocol (swallow capsules or to hold enema content for at least 15 minutes)
* Pregnancy
* Inability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessing restoration of the fecal microbiota after 14 day of H. pylori antibiotic regimen | 4 weeks
  A change of <10% of fecal microbial diversity before antibiotics and after FMT

SECONDARY OUTCOMES:
Side effects rate of auto-FMT delivered through capsules | 4 months
  Side effects will be recorded at every visit and will be compared between the groups
Side effects rate of auto-FMT delivered through enema | 4 months
  Side effects will be recorded at every visit and will be compared between the groups
H pylori re-infection rate after auto-FMT procedure | 4 weeks
  4 week after each auto-transplantation a breath test for H. Pylori will be performed to evaluate whether auto-FMT results in re-infection. Re-infection is expected to be lower than 10%
Fecal microbial diversity change in auto-FMT delivered through capsules 18 weeks post FMT compared to 4 weeks post FMT | 18 weeks
  The microbial composition and diversity analysis at week 18 will be compared to microbial composition analysis at week 4 in patients receiving FMT through capsules and is expected to be higher than 10% in the intervention group
Fecal microbial diversity change in auto-FMT delivered through enema 18 weeks post FMT compared to 4 weeks post FMT | 18 weeks
  The microbial composition and diversity analysis at week 18 will be compared to microbial composition analysis at week 4 in patients receiving FMT through enema and is expected to be higher than 10% in the intervention group

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No